CLINICAL TRIAL: NCT01365390
Title: To Evaluate Incidence of Acute Otitis Media in Children Aged < 6 Years in Five East European Countries
Brief Title: To Evaluate the Incidence of Acute Otitis Media in Children in Five East European Countries
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115356
Record Dates: First submitted 2011-05-31; First posted 2011-06-03 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-05

CONDITIONS: Infections, Streptococcal
Keywords: prospective; Incidence; otitis; observational; Epidemiological; retrospective
MeSH Terms: conditions — Streptococcal Infections; Otitis | interventions — Data Collection; Retrospective Studies; Longitudinal Studies

STUDY DESIGN:
Observational Model: Cohort

GROUPS / COHORTS (1):
- Cohort A: Subjects aged < 6 years who are registered in primary care clinics of any of the participating countries (Estonia, Lithuania, Poland, Romania and Slovenia).
  Interventions: Other: Data collection (Retrospective); Other: Data collection (Prospective)

INTERVENTIONS:
Other: Data collection (Retrospective) — For the retrospective part of the study, the parent(s)/ legally acceptable representative(s) of the subjects will be interviewed to collect information on factors potentially related to risk for middle ear diseases. The medical records of the subjects will also be reviewed and all acute otitis media related problems that occurred during the last year prior to enrolment (for subjects aged 1 to < 6 years) or since birth (for subjects aged < 1 year) will be recorded in the electronic case report form.
Other: Data collection (Prospective) — For the prospective part of the study, the enrolled subjects will be followed up for a period of 1 year starting from the consent date, during which the parent(s)/ legally acceptable representative(s) will be asked to bring the subject for a visit each time they notice symptoms of acute otitis media or respiratory tract infection in the subject. In case AOM is diagnosed by the investigator, detailed information on the signs, symptoms, severity, course and treatment will be recorded. The parent(s)/ legally acceptable representative(s) of the subjects will also be required to fill up a parental quality of life questionnaire and an Otitis Media-6 children's quality of life questionnaire.

SUMMARY:
The aim of this study is to provide baseline acute otitis media data in East European countries.

DETAILED DESCRIPTION:
Each subject's involvement in this study will include a retrospective and prospective part.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that parent(s)/ legally acceptable representative(s) can and will comply with the requirements of the protocol.
* A male or female subject aged < 6 years at the time of enrolment.
* The investigator has access to the medical records that contain the medical history of the subjects for one year prior to enrolment (for subjects aged 1 to < 6 years) or from birth (for subjects aged < 1 year).
* Written informed consent obtained from either both parents/ LARs or from one parent/ LAR of the subject with the declaration of cooperation for one year after enrolment.

Exclusion Criteria:

* Acute otitis media episode at the time of enrolment.
* Upper respiratory tract infection at the time of enrolment.

Max Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects aged < 6 years who are registered in primary care clinics of any of the participating countries (Estonia, Lithuania, Poland, Romania and Slovenia) will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 2258 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of acute otitis media in subjects aged < 6 years as diagnosed by a family physician and documented in medical records - retrospective part of the study | Retrospective data for 12 months prior to study entry for subjects aged > 1 year or for the entire period since birth for subjects aged < 1 year
Occurrence of acute otitis media in subjects aged < 6 years as diagnosed by the physician or specialist - prospective part of the study | Prospective data for 12 months after study entry

SECONDARY OUTCOMES:
Prevalence of otitis media with effusion among acute otitis media cases aged < 6 years in the four consecutive seasons of the year | Prospective data for 12 months after study entry
Occurrence of suspected acute otitis media as reported by the parent(s)/ legally acceptable representative(s) (and not diagnosed by any physician) during the bi-monthly follow-up | Prospective data for 12 months after study entry
Occurrence of recurrent acute otitis media | Retrospective data for 12 months prior to study entry for subjects aged > 1 year or for the entire period since birth for subjects aged < 1 year and prospective data for 12 months after study entry
Occurrence of acute otitis media treatment failures | Prospective data for 12 months after study entry
Assessment of the impact of acute otitis media on the quality of life of the subject and family by the parental quality of life questionnaire and the Otitis Media-6 children's quality of life questionnaire | Prospective data for 12 months after study entry
Direct medical, direct non-medical costs and indirect medical costs of one incident of acute otitis media | Prospective data for 12 months after study entry
Occurrence of acute otitis media as diagnosed by the study physician or any other doctor | Prospective data for 12 months after study entry
Use of antimicrobial therapy and other forms of treatment for acute otitis media, diagnostic procedures | Prospective data for 12 months after study entry

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (21):
- GSK Investigational Site, Tallinn, Estonia
- GSK Investigational Site, Vilnius, Lithuania
- Poland (10):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Kielce
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Tarnów
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wejherowo
  - GSK Investigational Site, Wola
  - GSK Investigational Site, Łęczna
- Romania (5):
  - GSK Investigational Site, Bacau
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Galati
- Slovenia (4):
  - GSK Investigational Site, Ljubljana
  - GSK Investigational Site, Maribor
  - GSK Investigational Site, Ptuj
  - GSK Investigational Site, Ruše

REFERENCES:
- [Derived] Usonis V, Jackowska T, Petraitiene S, Sapala A, Neculau A, Stryjewska I, Devadiga R, Tafalla M, Holl K. Incidence of acute otitis media in children below 6 years of age seen in medical practices in five East European countries. BMC Pediatr. 2016 Jul 26;16:108. doi: 10.1186/s12887-016-0638-2. PMID 27457584